CLINICAL TRIAL: NCT06776718
Title: Comparison of VNOTES and Vaginal Hysterectomy for Benign Indications
Brief Title: VNOTES and Vaginal Hysterectomy for Benign Indications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Mete Kırlangıç, Assoc Prof, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/514/214/25
Record Dates: First submitted 2024-12-24; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Hysterectomy; Hysterectomy, Benign Uterine Diseases; Hysterectomy, Vaginal
Keywords: vNOTES; vaginal hysterectomy; benign gynecology; surgical outcomes; Pain
MeSH Terms: conditions — Pain | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vNOTES hysterectomy for benign indications (Experimental)
  Interventions: Procedure: vNOTES
- Vaginal hysterectomy for benign indications (Experimental)
  Interventions: Procedure: vaginal hysterectomy

INTERVENTIONS:
Procedure: vNOTES — vNOTES for benign hysterectomy
  Arms: vNOTES hysterectomy for benign indications
Procedure: vaginal hysterectomy — vaginal hysterectomy for benign hysterectomy
  Arms: Vaginal hysterectomy for benign indications

SUMMARY:
This study aimed to compare the surgical outcomes of Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) and conventional vaginal hysterectomy (VH) for benign gynecological conditions.

A prospective analysis will conducted at a tertiary hospital from January 2025 to February 2025. Patients aged 40-80 who underwent hysterectomy for benign indications will included. Outcomes will assessed included surgical outcomes, Visual Analog Scale (VAS) pain scores, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* aged between 40 and 80 years
* undergo hysterectomy for benign gynecological conditions

Exclusion Criteria:

* history of urogynecological surgery (including pelvic organ prolapse surgery and mid-urethral sling procedures),
* suspected gynecologic malignancies,
* endometriosis,
* tubal-ovarian abscesses,
* pelvic organ prolapse exceeding grade 2,
* individuals who refused to participate in the study

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
the duration of surgery | The time from the beginning to the end of the operation
  İnterval from initial incision to the completion of vaginal cuff closure (minute)

SECONDARY OUTCOMES:
Hospitalization time | through study completion, an average of 1 month
  Time from surgery to discharge (hours)
VAS score | postoperative 6th and 24 th hour
  Visual Analog Score for pain at postoperative 6th and 24 th hour (0-10)
Uterin volume | through study completion, an average of 1 month
  Uterine volume is quantified in milimeters based on measurement of pathological specimens, calculate using the formula (Uterine volume (ml)= (anterior-posterior diameter)* (sagital diameter) * (transverse diameter) * 0,0005236
Re-admission | within 1 month after discharge
  Re-admission to hospital after discharge (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yildiz P, Keles E, Yildiz G, Birol Ilter P, Temocin RB, Kaya C, Mat E. Health-related quality of life following hysterectomy by vNOTES versus conventional laparoscopy. Minim Invasive Ther Allied Technol. 2024 Aug;33(4):232-236. doi: 10.1080/13645706.2024.2323100. Epub 2024 Mar 4. PMID 39084252
- [Background] Merlier M, Collinet P, Pierache A, Vandendriessche D, Delporte V, Rubod C, Cosson M, Giraudet G. Is V-NOTES Hysterectomy as Safe and Feasible as Outpatient Surgery Compared with Vaginal Hysterectomy? J Minim Invasive Gynecol. 2022 May;29(5):665-672. doi: 10.1016/j.jmig.2022.01.007. Epub 2022 Jan 21. PMID 35074513
- [Background] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol B, Bosteels J. Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery versus laparoscopy as a day-care procedure: a randomised controlled trial. BJOG. 2019 Jan;126(1):105-113. doi: 10.1111/1471-0528.15504. PMID 30325565
- [Background] Pickett CM, Seeratan DD, Mol BWJ, Nieboer TE, Johnson N, Bonestroo T, Aarts JW. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2023 Aug 29;8(8):CD003677. doi: 10.1002/14651858.CD003677.pub6. PMID 37642285